CLINICAL TRIAL: NCT03124537
Title: Increasing Physical Activity Among Sedentary Older Adults:What, Where, When, and With Whom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Margie Lachman, Professor of Psychology, Brandeis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Appstudy#16130; 5P30AG048785 (NIH)
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Sedentary Lifestyle; Self Efficacy; Control Locus; Aging
Keywords: Physical Exercise; Behavior Change
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Both conditions will receive the App for use on an iphone. The control group will just have the accelerometer program to set step goals and to count steps. The experimental condition will have the accelerometer to set goals and count steps in addition to the schedule, map and social components.
Who Masked: Participant
Masking Description: The participants are aware of the nature of the App features they are given. They are not aware of whether they are in an experimental or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Control Condition (Experimental): The control group will just have the App with the accelerometer program to set step goals and to count and record steps for 1 month
  Interventions: Behavioral: App Condition Control
- App Experimental condition (Experimental): The experimental condition will set step goals and have the schedule, map, and social components for 1 month.
  Interventions: Behavioral: App Experimental condition

INTERVENTIONS:
Behavioral: App Experimental condition — This group were given the app to 1) count their steps, 2) add walks to their daily schedules, 3) create maps of their walking routes, and 4) text friends to invite them for a walk. Participants are asked to set a daily step goal and they can see how many steps they've taken each day since using the app. 2) There is an interface where participants can create maps based on walking routes. 3) They will also have the option to use a daily schedule to plan certain times in the day that they can walk. 4) The social feature gives participants the option to message friends, co-workers, or neighbors in one's contact list to invite them for a walk. They were also asked to respond to two questions twice a day about their mood and energy levels.
  Arms: App Experimental condition
Behavioral: App Condition Control — This group received the app with the first component, the ability to count steps and set daily step goals. This group will also be able to track walks to see the time, distance, and steps of each walk, but not see these walks displayed as a map. This group will monitor their daily steps over a one-month period, and will be asked to use the app as much as possible. They were also asked to respond to two questions twice a day about their mood and energy levels.
  Arms: App Control Condition

SUMMARY:
The goal of this study is to develop a smart phone app to administer a behavior change program that helps adults to increase daily steps by planning where, when, and with whom to walk. The investigators tested the effectiveness of the walking program app for increasing the number of daily steps among sedentary older adults. The investigators examined the effects on self-efficacy and social integration/support.

DETAILED DESCRIPTION:
Physical activity is broadly beneficial for physical, psychological, and cognitive aspects of health, yet only one in five U.S. adults meets the CDC physical activity guidelines. Making physical activity accessible and feasible throughout life is an important public health policy objective that is within reach with the right kind of behavioral and environmental supports. The project aims to provide such supports for an active lifestyle thereby contributing to healthy aging. The goal of this project is to increase physical activity (i.e., walking) in sedentary older adults by providing the environmental and behavioral resources to incorporate additional steps into their daily lives. The investigators used a behavioral approach that fosters a sense of control and facilitates planning by focusing on the what, when, where, and with whom aspects of their physical activity. The investigators proposed a user-friendly, practical way to increase steps. By providing people with specific, tailored information about the number of steps one can get by walking a certain distance or during a certain amount of time, participants can better plan when, where, and with whom they will be able to achieve the desired number of steps, break goals into manageable portions (at different times throughout the day or week), and thereby increase the likelihood of goal achievement.

During the app development phase, the investigators demonstrated the app to 10 older adults to get their input. The goal was to get their feedback about the app features and to make sure it is user friendly. The investigators asked questions about the ease of using the app and their understanding of the app features. The interviewer recorded their answers to share with the research team and app developer. Modifications to the app were made based on the feedback.

During the next phase of the study, the investigators tested whether the full app program was successful in increasing steps and whether it was more effective than the basic app that only includes step counting and goals, similar to a fitness tracker or pedometer. Sixty participants were randomly assigned to two conditions: the app with step counting and goals alone (control), or the full version of the app with the step counting and goals, schedule, maps, and social components (experimental). It was predicted that the intervention group would improve more on outcome measures than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary adults, who own an iphone with step-tracking capabilities (5s or later).
* Participants must be fit enough to walk for at least 20 minutes at a time.

Exclusion Criteria:

* Cognitive impairment
* A recent (within the past 6 months) cardiovascular event, or fall.
* A doctor has advised them not to walk
* Anyone who already exercises regularly: walks for exercise more than 30 minutes per day, or does other forms of exercise 150 minutes per week or more, will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margie Lachman, Ph.D., Principal Investigator — Brandeis University
Locations (1):
- Brandeis University, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sullivan AN, Lachman ME. Behavior Change with Fitness Technology in Sedentary Adults: A Review of the Evidence for Increasing Physical Activity. Front Public Health. 2017 Jan 11;4:289. doi: 10.3389/fpubh.2016.00289. eCollection 2016. PMID 28123997
- [Derived] Bisson AN, Sorrentino V, Lachman ME. Walking and Daily Affect Among Sedentary Older Adults Measured Using the StepMATE App: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Dec 1;9(12):e27208. doi: 10.2196/27208. PMID 34855609

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | App Control Condition | App Experimental Condition
Started | 41 | 45
Completed | 31 | 32
Not Completed | 10 | 13
Not completed — Lost to Follow-up | 3 | 5
Not completed — App Crash, Incomplete Data | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | App Control Condition | App Experimental Condition | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.71 (6.30) | 63.63 (7.89) | 64.16 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 30 | 32 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 28 | 28 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Steps Walked
Description: Number of steps recorded daily on the phone app, weekly step averages
Time Frame: Daily for one month
Population: Participants were excluded if they dropped out of the study or experienced the app crash. Analyses were conducted using an intent to treat population. Daily step averages less than 500 steps were classified as a missing day of data. Weekly step averages were only calculated if there were 4 or more days of valid data.
Measure: Mean (Standard Deviation); unit: Average Daily Steps
Arm/Group | App Control Condition | App Experimental Condition
Number analyzed (Participants) | 31 | 32
Average Daily Steps
  Baseline Steps: number analyzed (Participants) | 26 | 26
  Baseline Steps | 3910.37 (2971.40) | 3477.66 (1749.29)
  Week 1 Steps: number analyzed (Participants) | 30 | 30
  Week 1 Steps | 5744.00 (2398.89) | 5279.66 (2445.76)
  Week 2 Steps: number analyzed (Participants) | 30 | 31
  Week 2 Steps | 5317.08 (2249.66) | 5116.88 (2983.89)
  Week 3 Steps: number analyzed (Participants) | 30 | 30
  Week 3 Steps | 5858.90 (2446.95) | 5197.21 (2968.79)
  Week 4 Steps: number analyzed (Participants) | 30 | 31
  Week 4 Steps | 5155.42 (2505.59) | 5285.26 (3493.65)
Statistical Analysis 1: Comparison: App Control Condition vs App Experimental Condition; Tested whether weekly steps increased from the baseline week in both conditions (main effect of time); Test type: Superiority; p < .001, Mixed Models Analysis; Controlling for age, sex, condition, education, and health
Statistical Analysis 2: Comparison: App Control Condition vs App Experimental Condition; Tested whether weekly step increases from the baseline week differed between the two conditions (time by condition interaction); Test type: Superiority; p = .846, Mixed Models Analysis — Controlling for age, sex, education, and health

2. Secondary Outcome: Exercise Self-efficacy
Description: A modified version of Bandura's Exercise Self-Efficacy scale (Bandura, 1997) was used in the current study. This 9-item scale assesses how sure one is that they would exercise under different conditions or constraints (e.g. How sure are you that you will exercise when you are feeling down or depressed?), with answer choices ranging from not sure at all (1) to very sure (4). The 9 items are averaged to create a composite score, where a higher score indicates greater exercise self-efficacy (Neupert et al., 2009).
Time Frame: Baseline and one month from the start of the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Control Condition | App Experimental Condition
Number analyzed (Participants) | 31 | 32
units on a scale
  Pre-test | 2.61 (0.67) | 2.88 (0.83)
  Post-test | 2.43 (0.83) | 2.54 (0.92)
Statistical Analysis 1: Comparison: App Control Condition vs App Experimental Condition; Tested whether exercise self-efficacy increased from the baseline week to the end of the intervention in both conditions (main effect of time); Test type: Superiority; p = .571, Mixed Models Analysis — Controlling for age, sex, condition, education, and health
Statistical Analysis 2: Comparison: App Control Condition vs App Experimental Condition; Tested whether exercise self efficacy increases from the baseline to the end of the intervention differed between the two conditions (time by condition interaction); Test type: Superiority; p = .361, Mixed Models Analysis; Controlling for age, sex, education, and health

3. Secondary Outcome: Exercise Control Beliefs
Description: Control over exercise was measured using the 6-item Exercise Control Beliefs Scale (Neupert, Lachman, & Whitbourne, 2009). Items assess the beliefs about one's control over exercise (e.g., I am confident in my ability to do an exercise routine), with answer choices ranging from strongly disagree (1) to strongly agree (5). The 6 items are averaged to create a mean exercise control score, with a higher score indicating greater control over exercise.
Time Frame: Baseline and one month from the start of the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Control Condition | App Experimental Condition
Number analyzed (Participants) | 31 | 32
units on a scale
  Pre-test | 4.39 (0.48) | 4.23 (0.53)
  Post-test | 4.31 (0.51) | 4.25 (0.62)
Statistical Analysis 1: Comparison: App Control Condition vs App Experimental Condition; Tested whether exercise control increased from the baseline week to the end of the intervention in both conditions (main effect of time); Test type: Superiority; p = .564, Mixed Models Analysis; Controlling for age, sex, condition, education, and health
Statistical Analysis 2: Comparison: App Control Condition vs App Experimental Condition; Tested whether exercise control belief increases from the baseline to the end of the intervention differed between the two conditions (time by condition interaction); Test type: Superiority; p = .641, Mixed Models Analysis; Controlling for age, sex, education, and health

4. Secondary Outcome: Social Contact Through the App
Description: Number of participants who sent at least one text message via the app
Time Frame: During the one month intervention
Measure: Number; unit: participants
Arm/Group | App Control Condition | App Experimental Condition
Number analyzed (Participants) | 31 | 32
participants | 0 | 1

5. Secondary Outcome: Daily Mood and Energy Levels
Description: Twice at random times, each day, mood and energy levels were assessed. A popup notification asked participants to rate their current mood (unhappy, neutral, happy) and energy (low, neutral, high) on a slider scale. Scores were converted by the StepMATE app to a 0-10 scale, with 0 indicating low mood/energy, and 10 indicating high mood/energy. If both mood and energy assessments were completed in one day, they were averaged to create daily average scores, one for mood and one for energy. Data presented below are the average of all daily scores across the month, while daily averages were used in the analyses.
Time Frame: Daily
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Control Condition | App Experimental Condition
Number analyzed (Participants) | 31 | 32
units on a scale
  Mood | 6.91 (1.67) | 6.53 (1.35)
  Energy | 5.58 (1.35) | 5.80 (1.61)
Statistical Analysis 1: Comparison: App Control Condition vs App Experimental Condition; Tested whether daily walking was related to mood within-persons; Test type: Superiority; p < .001, Mixed Models Analysis; Controlling for age, sex, condition, education, health, and average steps
Statistical Analysis 2: Comparison: App Control Condition vs App Experimental Condition; Tested whether daily walking was related to energy within-persons; Test type: Superiority; p = .003, Mixed Models Analysis; Controlling for age, condition, education, health, and average steps
Statistical Analysis 3: Comparison: App Control Condition vs App Experimental Condition; Tested whether the relationship between daily walking and mood differed between males and females (steps by sex interaction); Test type: Superiority; p < .001, Mixed Models Analysis; Controlling for age, sex, condition, education, health, and average steps
Statistical Analysis 4: Comparison: App Control Condition vs App Experimental Condition; Tested whether the relationship between daily walking and energy differed between males and females (steps by sex interaction); Test type: Superiority; p < .001, Mixed Models Analysis; Controlling for age, condition, education, health, and average steps

6. Secondary Outcome: Self-Reported Vigorous Physical Activity
Description: Vigorous PA was measured using the question 'How often do you engage in vigorous physical activity that causes your heart to beat so rapidly that you can feel it in your chest and you perform the activity long enough to work up a good sweat and are breathing heavily?', with answer choices ranging from never (0) to several times a week (5).
Time Frame: Baseline and one month from the start of the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Control Condition | App Experimental Condition
Number analyzed (Participants) | 31 | 32
units on a scale
  Pre-test | 1.94 (1.83) | 2.13 (1.83)
  Post-test | 2.77 (1.63) | 2.53 (1.83)
Statistical Analysis 1: Comparison: App Control Condition vs App Experimental Condition; Tested whether self-reported vigorous physical activity increased from the baseline week to the end of the intervention in both conditions (main effect of time); Test type: Superiority; p = .011, Mixed Models Analysis; Controlling for age, sex, condition, education, and health
Statistical Analysis 2: Comparison: App Control Condition vs App Experimental Condition; Tested whether self-reported vigorous physical activity increases from the baseline to the end of the intervention differed between the two conditions (time by condition interaction); Test type: Superiority; p = .232, Mixed Models Analysis; Controlling for age, sex, education, and health

7. Secondary Outcome: Self-Reported Moderate Physical Activity
Description: Moderate PA was measured with the question 'How often do you engage in moderate physical activity that is not physically exhausting, but it causes your heart rate to increase slightly and you typically work up a sweat?', with answer choices ranging from never (0) to several times a week (5).
Time Frame: Baseline and one month from the start of the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Control Condition | App Experimental Condition
Number analyzed (Participants) | 31 | 32
units on a scale
  Pre-Test | 3.94 (1.44) | 3.50 (1.67)
  Post-test | 4.13 (1.18) | 3.63 (1.76)
Statistical Analysis 1: Comparison: App Control Condition vs App Experimental Condition; Tested whether self-reported moderate physical activity increased from the baseline week to the end of the intervention in both conditions (main effect of time); Test type: Superiority; p = .530, Mixed Models Analysis; Controlling for age, sex, condition, education, and health
Statistical Analysis 2: Comparison: App Control Condition vs App Experimental Condition; Tested whether self-reported moderate physical activity increases from the baseline to the end of the intervention differed between the two conditions (time by condition interaction); Test type: Superiority; p = .831, Mixed Models Analysis; Controlling for age, sex, education, and health

8. Secondary Outcome: Self-Reported Light Physical Activity
Description: Light PA was measured using the question 'How often do you engage in light physical activity that requires little physical effort?', with answer choices ranging from never (0) to several times a week (5).
Time Frame: Baseline and one month from the start of the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Control Condition | App Experimental Condition
Number analyzed (Participants) | 31 | 32
units on a scale
  Pre-test | 4.77 (0.56) | 4.69 (0.64)
  Post-test | 4.61 (0.84) | 4.78 (0.61)
Statistical Analysis 1: Comparison: App Control Condition vs App Experimental Condition; Tested whether self-reported light physical activity increased from the baseline week to the end of the intervention in both conditions (main effect of time); Test type: Superiority; p = .199, Mixed Models Analysis; Controlling for age, sex, condition, education, and health
Statistical Analysis 2: Comparison: App Control Condition vs App Experimental Condition; Tested whether self-reported light physical activity increases from the baseline to the end of the intervention differed between the two conditions (time by condition interaction); Test type: Superiority; p = .203, Mixed Models Analysis; Controlling for age, sex, education, and health

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | App Control Condition | App Experimental Condition
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/45
Other Adverse Events (participants affected / at risk) | 0/41 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT03124537/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT03124537/ICF_001.pdf